CLINICAL TRIAL: NCT06405581
Title: The Impact of Frailty on Cardiopulmonary Resuscitation Adverse Outcomes in Patients Requiring Code Blue Activation
Status: Recruiting | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zeliha Alicikus, Head of Anesthesiology and Reanimation department,Assoc Prof, Umraniye Education and Research Hospital
Other Study IDs: UERH-AR-ZT-05
Record Dates: First submitted 2023-12-29; First posted 2024-05-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Arrest; Frailty; Respiratory Arrest
MeSH Terms: conditions — Heart Arrest; Frailty; Apnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Edmonton frailty scale ≥ 7: The frailty status of the patients will be assessed using the Edmonton frailty scale.
  According to the Edmonton frailty scale;
  * (0-5): not frail
  * (6-7): sensitive
  * (8-9): slightly fragile
  * (10-11): moderately fragile,
  * (12-17): extremely fragile
  Interventions: Other: Edmonton frailty scale calculation
- Edmonton frailty scale below 7: The frailty status of the patients will be assessed using the Edmonton frailty scale.
  According to the Edmonton frailty scale;
  * (0-5): not frail
  * (6-7): sensitive
  * (8-9): slightly fragile
  * (10-11): moderately fragile,
  * (12-17): extremely fragile
  Interventions: Other: Edmonton frailty scale calculation

INTERVENTIONS:
Other: Edmonton frailty scale calculation — The frailty status of the patients will be assessed using the Edmonton frailty scale.
  According to the Edmonton frailty scale;
  * (0-5): not frail
  * (6-7): sensitive
  * (8-9): slightly fragile
  * (10-11): moderately fragile,
  * (12-17): extremely fragile

SUMMARY:
The aim of this study was to determine the independent association of frailty with cardiopulmonary resuscitation and predictive factors in patients triggering code blue response

DETAILED DESCRIPTION:
Out-of-hospital cardiac arrest remains an important cause of death in developed countries with an average adult survival rate of 5.6% . In contrast, in-hospital cardiac arrests have been reported to have a survival rate between 4.1% and 40% and several factors have been shown to affect survival rates. These factors include patient and physiologic factors such as age, initial rhythm disturbance and duration of cardiopulmonary resuscitation (CPR), as well as hospital and logistic factors such as location and timing of the arrest.Code blue (CC) is the emergency call and management systems for respiratory or cardiac arrest. CC is used worldwide for the same emergency and the same color. The CC is the organization that initiates certain systems to initiate, perform and terminate the intervention of the designated responsible team. CC is given by a doctor (emergency, anesthesia and reanimation, internal medicine, pediatrics, intensive care specialist), anesthesia technician, nurse. The CC team is a team that prevents clinical death quickly, effectively and safely to provide life-saving support to patients. The CC team provides immediate intervention to patients, their relatives and all hospital staff. While the prevalence of frailty is 10-25% in the elderly aged 65 years and over, it increases to 30-45% in those aged 85 years and over. There are no definitive data on the prevalence of frail elderly in Turkey. The definition of frail elderly syndrome emerged as a concept in geriatrics and gerontology in the 1980s in response to the growing need for a unifying diagnosis among seemingly disparate and nonspecific disease presentations in older adults. The main symptoms are weight loss, weakness, fatigue and immobility, while the main findings are sarcopenia, osteopenia, malnutrition, impaired balance and gait, and slow walking. The importance of the definition of frailty comes from the fact that it is an alarm table used to indicate the susceptibility of the elderly to conditions such as clinical deterioration, falls and mortality over time. Frailty is a syndrome that can be prevented or at least postponed if diagnosed at an early stage. In fact, the frail elderly constitute a group vulnerable to adverse events with poor prognosis Mortality and complication rates are higher in elderly surgical patients than in younger surgical patients. Surgical risk is even higher in frail elderly patients. Regardless of the type of surgery and whatever assessment tool is used, the presence of frailty is associated with an approximately two- to threefold increased risk of adverse surgical outcome. Numerous studies have shown that frailty is a risk factor for postoperative complications, longer hospital stay and loss of functional independence at discharge. Therefore, identifying older patients with frailty offers opportunities to provide improved risk stratification and targeted interventions to improve outcomes The Edmonton Frailty Scale, a performance-based multidimensional frailty assessment tool, was designed by non-geriatricians in the west to help assess and screen frail older patients in primary care and at the bedside. It consists of 11 questions relating to nine different domains such as awareness, social support, mood, nutrition and functional performance. The result correlates well with the clinical impression of geriatricians through detailed history and physical examination.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients

Exclusion Criteria:

* pregnant patients

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with hospitalization and those who are not inpatients (in the outpatient clinic system) requiring Code Blue will be included in the study.
Sampling Method: Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
code blue reason | years
  comorbid disease and dog usage
duration of CPR time | hours
  between the time of giving the blue code and the end of CPR

SECONDARY OUTCOMES:
the airway equipment used | days
  intubation, supraglottic airway devices, tracheostomy, cricothyroidectomy, fiberbronchoscopy
mortality and morbidity | mounts
  presence and duration of intensive care unit stay

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Education and Research Hospital, Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No